CLINICAL TRIAL: NCT01422109
Title: Comparative Pharmacokinetics After Single Oral Administration of YH14659, a Fixed Dose Combination Versus Coadministration of Separate Constituents in Healthy Male Volunteers
Brief Title: Comparative Pharmacokinetics of YH14659
Acronym: YH14659
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YH14659-101
Record Dates: First submitted 2011-08-16; First posted 2011-08-23 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Acute Coronary Syndrome
Keywords: YH14659; Aspirin; Clopidogrel; Yuhan
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: YH14659
- Group B (Active Comparator)
  Interventions: Drug: clopidogrel & aspirin

INTERVENTIONS:
Drug: YH14659 — YH14659 capsule by oral
  Arms: Group A
Drug: clopidogrel & aspirin — clopidogrel tablet(75mg) + aspirin capsules(100mg) by oral
  Arms: Group B

SUMMARY:
The objective of this study is to compare pharmacokinetics after single oral administration of 2 capsules of YH14659, a fixed-dose combination of clopidogrel and aspirin developed by Yuhan Corporation versus co-administration of Plavix (clopidogrel) and Astrix (aspirin) in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* The patient or legally authorized representative must sign a written informed consent, prior to the any procedure, using a form that is approved by the local Institutional Review Board after detail explanation of the purpose, contents, and characteristic of the drug
* Healthy male volunteers of aged between 20 years to 55 years
* Have standard weight of ≤ ±20% based on Broca index* (Broca index: ideal weight(kg) = (height(cm)-100) x 0.9)
* Have no history of neither congenital nor chronic disease
* Have no history of abnormal symptoms or opinions as a result of physical examination (medical checkup)
* Eligible subjects with acceptable medical history, physical examination laboratory tests, ECG during screening period

Exclusion Criteria:

* Received any drug that induce or/and inhibit drug metabolizing enzyme such as barbital within the last 28 days prior to the first administration
* Shown symptoms doubtful as an acute disease within the last 28 days prior to the first administration
* Have signs of bleeding symptoms or/and history of disease such as: gum bleeding, hard to control hemorrhage, easily suffer from bruise, and etc.
* Have disease that can affect absorption, distribution, metabolism and excretion of the drug such as: inflammatory bowel disease, gastric ulcer, duodenal ulcer, hepatic disorders, and gastrointestinal tract surgery except appendectomy
* Have a known allergy(except mild allergic rhinitis which does not require treatment) or hypersensitivity to drugs
* Have the following abnormal findings on diagnosis;

  * have AST or ALT > 1.25 times of normal upper limit
  * have total bilirubin > 1.5 times of normal upper limit
  * have higher PT, aPPT, BT than normal range
  * have PLT below 150,000 or above 350,000
* Have been drug abuse, excessive caffeine (> 5 cups/day), heavy smoking (>10 cigarettes/day), continuous alcohol intake (> 30g/day) or have drunk within the last 7 days prior to the first administration
* Have been on a diet that can affect absorption, distribution, metabolism and excretion of the drug (especially grapefruit juice 7 days prior to the first administration)
* Donated blood within 60 days prior to the first administration
* Participated in any other clinical trials within 60 days prior to the first administration
* Have used any drug which is thought to affect this study by principal investigator 10 days prior to the first administration
* Subject who is judged to be ineligible by principal investigator or sub-investigator

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration(Cmax) of clopidogrel | 14 days
Area under the time-concentration curve to last concentration(AUCt) of clopidogrel | 14 days
Maximum plasma concentration(Cmax) of acetylsalicylic acid | 14 days
Area under the time-concentration curve to last concentration(AUCt) of acetylsalicylic acid | 14 days

SECONDARY OUTCOMES:
Cmax of salicylic acid, the major active metabolite of aspirin | 14 days
AUCt of salicylic acid, the major active metabolite of aspirin | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, MD, PhD., Principal Investigator — Inje University
Locations (1):
- Yuhan Corporation, Seoul, South Korea